CLINICAL TRIAL: NCT04254939
Title: A Phase I/II Clinical Study of Avapritinib in Chinese Subjects With Unresectable or Metastatic Gastrointestinal Stromal Tumor
Brief Title: A Study of CS3007 in Subjects With Gastrointestinal Stromal Tumor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Collaborators: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS3007-101
Record Dates: First submitted 2019-12-09; First posted 2020-02-05 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — avapritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CS3007(BLU-285) (Experimental)
  Interventions: Drug: CS3007 (BLU-285)

INTERVENTIONS:
Drug: CS3007 (BLU-285) — A modified "3+3" dose escalation design will be adopted. Each group will enroll 3-6 subjects. Avapritinib will be administered orally at the starting of 200 mg QD. A cycle consists of 28 consecutive days.

SUMMARY:
This study is an open-label, multicenter, phase I/II study to evaluate the safety, PK and clinical efficacy of avapritinib in Chinese subjects with unresectable or metastatic GIST. The study consists of two parts: dose escalation (phase I) and dose expansion (phase II).

ELIGIBILITY:
Inclusion criteria:

1. For phase I study, the subject must have histologically or cytologically confirmed unresectable or metastatic GIST that progressed after imatinib and at least one additional TKI treatment, or who cannot tolerate the standard treatment or have D842V mutation in the PDGFRα gene.
2. For phase II study:

   i) Group 1: Chinese subjects with unresectable GIST harboring D842V mutation in PDGFRα gene.

   ii) Group 2: Chinese third-line and fourth-line or later subjects with unresectable GIST that has progressed after standard treatment and/or do not tolerate standard treatment, and do not have a known D842V mutation in the PDGFRα gene.
3. Subjects with at least one measurable lesion as defined per mRECIST v1.1
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.

Exclusion Criteria

1. Subject has any of the laboratory results that meet exclusion criteria
2. Subjects who have previously received antineoplastic medication, including Chinese herbal drugs or Chinese medicine products with antineoplastic indications, for less than 5 half-lives or 14 days, whichever is shorter, prior to the first dose of the investigational product.
3. The subject received neutrophil growth factor support within 14 days prior to the first dose of investigational product.
4. Subjects received treatment with a strong inhibitor or strong or moderate inducer of cytochrome P450 (CYP) 3A4 within 14 days prior to the first dose of study drug, or requires continuous intake of above medications or foods during study period.
5. Subject received a major surgery (not including minor procedures, e.g., central venous catheterization, tumor needle biopsy, feeding tube placement) within 14 days prior to the first dose of investigational product.
6. Diagnosis of any other malignancy within 1 year prior to the first dose of investigational product or the subject is under treatment for another malignancy.
7. Corrected QT interval > 450 msec calculated using Fridericia's formula.
8. Subject has history of seizure (e.g. epilepsy) or requires antiepileptic medication treatment.
9. History of cerebrovascular accident or transient ischemic attack within one year prior to the first dose of the investigational product.
10. Known risk of intracranial hemorrhage, e.g., history of cerebral aneurysm or subdural or subarachnoid hemorrhage.
11. With primary brain malignancy or brain metastasis.
12. With clinically significant, uncontrolled cardiovascular disease, including congestive heart failure of New York Heart Association (NYHA) class II, III or IV, myocardial infarction or unstable angina in the past 6 months, or uncontrolled hypertension.
13. Unwilling or unable to comply with scheduled visits, treatment plan, laboratory tests or other study procedures/restrictions.
14. With previous or current clinically significant disorder, medical condition, history of surgery, physical issue or laboratory finding, which, in the investigator's judgment, might affect the subject's safety, change the absorption, distribution, metabolism or excretion of the investigational product, or interfere with the evaluation of study result.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Phase I: Recommended Phase II dose (RP2D), incidence of dose limiting toxicities (DLT) in Cycle 1, incidence and severity of adverse events and serious adverse events and changes in vital signs, clinical laboratory results and ECG findings | at the end of Cycle 1 (each cycle is 28 days) for RP2D and DLT; during every cycle through 30 days after the last dose of study drug, an average of approximately 24 months, for other measures
Phase II: ORR based on mRESIST 1.1 | At Cycle 3 (each cycle is 28 days) Day 1, then every 2 cycles until Cycle 13, they every 3 cycles through study completion, disease progression or patient discontinuation from the study (whichever comes first), an average of approximately 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lin SHEN, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (16):
- China (16):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Wuhan Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang Medical University, Nanchang, Jiangxi
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Fudan University Zhongshan Hospital (General Surgery Department), Shanghai, Shanghai Municipality
  - Fudan University Zhongshan Hospital (Internal Tumor Department), Shanghai, Shanghai Municipality
  - Renji Hospital affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Xinjiang Medical University Cancer Hospital, Ürümqi, Xinjiang
  - The First Affiliated Hospital Zhe Jiang University, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Li J, Zhang X, Deng Y, Wu X, Zheng Z, Zhou Y, Cai S, Zhang Y, Zhang J, Tao K, Cui Y, Cao H, Shen K, Yu J, Zhou Y, Ren W, Qu C, Zhao W, Hu J, Wang W, Yang J, Shen L. Efficacy and Safety of Avapritinib in Treating Unresectable or Metastatic Gastrointestinal Stromal Tumors: A Phase I/II, Open-Label, Multicenter Study. Oncologist. 2023 Feb 8;28(2):187-e114. doi: 10.1093/oncolo/oyac242. PMID 36477870